CLINICAL TRIAL: NCT06897176
Title: Effects of Cerebrolysin on Language Ability in Non-fluent Aphasia Patients After Stroke: A Randomized, Placebo-controlled, Double-blinded, Single Center Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4-2024-0028
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Cerebrolysin Treatment) (Experimental): This group receives standard language therapy along with Cerebrolysin to improve language abilities in patients with non-fluent aphasia following a stroke. The treatment is evaluated through language assessment and neuroprotective effects.
  Interventions: Drug: Cerebrolyisin
- Placebo Group (Placebo Treatment) (Placebo Comparator): This group receives standard language therapy along with a placebo instead of Cerebrolysin. The placebo treatment is used to compare the effects of Cerebrolysin on language abilities and neuroprotection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cerebrolyisin — This intervention uses Cerebrolysin, which is a treatment aimed at improving language abilities and providing neuroprotection for patients with non-fluent aphasia following a stroke. Cerebrolysin is administered via intravenous injection, with the goal of improving language skills and promoting brain function recovery. The treatment is evaluated based on improvements in language abilities, neurological function recovery, and safety.
  Arms: Experimental Group (Cerebrolysin Treatment)
Drug: Placebo — The placebo is administered alongside standard language therapy to the patients with non-fluent aphasia following a stroke. This allows for comparison with the Cerebrolysin group to assess the impact of the treatment on language abilities and neurological function recovery. The goal is to evaluate the improvements in language skills, neurological function recovery, and safety, comparing the effects between the active treatment and placebo.
  Arms: Placebo Group (Placebo Treatment)

SUMMARY:
" This study aims to measure changes in language ability after adding cerebrolysin to standard treatment for non-fluent aphasia patients with post-stroke language impairment. The patients are divided into two groups: the experimental group, which receives a combination of standard treatment (speech therapy) and cerebrolysin, and the control group, which only receives standard treatment (speech therapy). By comparing the PK-WAB scores before and after drug administration, the study seeks to analyze the impact of cerebrolysin on language improvement. According to various stroke registries, 15-42% of patients in the subacute phase of stroke and 25-50% of patients with chronic stroke show symptoms of aphasia. Language therapy for stroke-related aphasia has become increasingly important due to its association with prolonged hospitalization, increased healthcare costs, mortality, and other negative prognostic factors .

After central nervous system damage such as stroke and traumatic brain injury, the administration of growth hormones and neurotrophic factors such as brain-derived neurotrophic factor (BDNF), glial cell line-derived neurotrophic factor (GDNF), nerve growth factor (NGF), and ciliary neurotrophic factor (CNTF) has been reported to influence nerve regeneration.

Cerebrolysin (EVER Neuro Pharma GmbH, AUSTRIA) is a multi-modal drug composed of low-molecular peptides and amino acids, which shows neuroprotective and neurotrophic effects similar to endogenous neurotrophic factors. Analysis of cerebrolysin using ELISA revealed that it contains CNTF, GDNF, IGF1, IGF2, and other factors structurally and functionally similar to neurotrophic factors (NTFs). Cerebrolysin activates the same PI3K/Akt pathway as BDNF, playing a crucial role in the growth, proliferation, differentiation, and migration of nerve cells, and promoting the maintenance, protection, and repair of neural networks. Additionally, it activates the SHH pathway, facilitating neuroplasticity and neurogenesis, thereby aiding the brain's self-repair process and functional recovery. Recent studies have shown that cerebrolysin reduces inflammation in the cerebral vasculature and improves the integrity of the blood-brain barrier by increasing tight junctions.

Cerebrolysin has shown excellent effects on motor function improvement in moderate-to-severe stroke patients in studies by Muresanu et al. 2016. and Chang et al. 2016. Based on these results, cerebrolysin has been included in stroke rehabilitation guidelines in Austria (2018), Germany (2020), Canada (2020), the European Neuroscience Society (2021), and the Korean Brain and Neurorehabilitation Society (2022). Furthermore, cerebrolysin has been included in the Canadian TBI guidelines for improving attention in patients with moderate-to-severe traumatic brain injury, and it is expected to be beneficial in the rehabilitation of both stroke and traumatic brain injury patients.

Although there is strong evidence that cerebrolysin improves motor function, attention, and consciousness levels after stroke or brain injury, its effect on language abilities remains unclear. Moreover, previous studies have limitations, including the use of the Western Aphasia Battery Test and heterogeneity in language assessments. Therefore, this study plans to conduct additional research using a well-designed, double-blind, placebo-controlled, randomized study to assess the effect of cerebrolysin on non-fluent aphasia, using a variety of evaluation tools to accurately measure improvements in language abilities."

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a first-episodic of ischemic or hemorrhagic stroke
2. Patients with lesions in the left supratentorial area confirmed by CT or MRI
3. Subacute phase within one month of stroke onset
4. Aged between 19 and 90 years
5. Patients diagnosed with non-fluent aphasia through the Korean version of the Western Aphasia Battery
6. Right-handed individuals assessed by the Edinburgh Handedness Inventory
7. Individuals who voluntarily provided written consent for participation in the clinical trial, either personally or through their legal representative
8. Native speakers of Korean

Exclusion Criteria:

1. Individuals with contraindications, including allergies to cerebrolysin
2. Multiple previous episode of stroke that had been managed.
3. Presence of significant pre-existing neurogenic disorders
4. Presence of significant psychiatric disorders such as major depressive disorder, schizophrenia, bipolar disorder, or dementia
5. History of alcohol or other substance abuse within 3 years of onset
6. Presence of severe liver, kidney, heart, or respiratory diseases
7. Medical findings from diagnostic tests indicating any of the following conditions (Total serum bilirubin > 4mg/dL, alkaline phosphatase > 250 U/L, SGOT/AST > 150 U/L. SGPT/ALT > 150 U/L., or creatinine >3.5 mg/dL)
8. Presence of an underlying medical condition with a life expectancy of less than 1 year
9. Pregnant or breastfeeding individuals
10. Participation in another therapeutic study

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-06-14 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Paradise Korean Western Aphasia Battery (PK-WAB) | up to 1 day
  It is a test used to evaluate the communication function of patients who have developed acquired neurological disorders, such as stroke, traumatic brain injury, and dementia. The test is divided into various language areas, including spontaneous speech, comprehension, repetition, naming, reading, and writing. Through the scoring of each item, the aphasia index and language index can be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Department and Research Institute of Rehabilitation Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No